CLINICAL TRIAL: NCT05157295
Title: Comparing Number of Injection Sites of In-office Intravesical Onabotulinumtoxin A Treatments for Overactive Bladder: A Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1791493
Record Dates: First submitted 2021-11-23; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Overactive Bladder Syndrome; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: One group of participants will receive the "experimental" treatment, which is 4 injections, and the other group of participants will receive the "standard" treatment, which is 20 injections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Group (Experimental): 100 U of onabotulinumtoxinA toxin diluted in 10 mL of saline cystoscopically injected into approximately 4 different detrusor muscle sites along the posterior bladder wall and dome.
  Interventions: Drug: OnabotulinumtoxinA
- Control Group (Active Comparator): 100 U of onabotulinumtoxinA toxin diluted in 10 mL of saline cystoscopically injected into approximately 20 different detrusor muscle sites along the posterior bladder wall and dome.
  Interventions: Drug: OnabotulinumtoxinA

INTERVENTIONS:
Drug: OnabotulinumtoxinA — 100 U of Onabotulinumtoxin A diluted in 10 mL of saline injected into the wall of the detrusor muscle at various sites

SUMMARY:
Overactive bladder (OAB) is a syndrome characterized by urinary urgency, with or without urinary incontinence, nocturia, and urinary frequency. Intravesical injection of onabotulinumtoxinA is approved by the US Food and Drug Administration for treatment of neurogenic and idiopathic OAB. Current standard of practice involves 100 U of onabotulinumtoxinA diluted in 10 ml saline cystoscopically injected into approximately 20 different detrusor muscle sites equally distributed along the posterior bladder wall and dome. This treatment was classically done in the operating room under general anesthesia, but now is typically performed in an office setting using local anesthesia (lidocaine) as this is more feasible and tolerable. Patients can experience discomfort and pain with each injection. Evidence has also shown that administering the same dose of onabotulinumtoxinA into fewer injection sites in the detrusor muscle (ranging from 3 to 10) results in equivalent efficacy compared to the current standard. However, it has yet to be determined if there is a significant difference in patient satisfaction and tolerability when the procedure is administered in an office setting using the same dosage with fewer injections. Our study aims to assess whether patient tolerance and satisfaction of intravesicular onabotulinumtoxinA increases with the use of 4 detrusor injections as opposed to 20 injections when performed in an office setting on women with OAB.

ELIGIBILITY:
Inclusion Criteria:

* females, adults 18 years of age and older, diagnosed with OAB

Exclusion Criteria:

* bladder pathology including nephrolithiasis, active urinary tract infection, bladder trauma, neurogenic bladder, patients who have previously received intravesical onabotulinumtoxin A injections, pregnant patients, minor patients, male patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Perceived pain of each participant before, during, and after the procedure on a scale of 0-10 | within the hour prior to initiating the intervention, and immediately at the conclusion of the 30-minute intervention
  The Pain Survey is a self-reported instrument used to assess pain before, during, and after a procedure. Possible scores range from 0 (no pain) to 10 (worst pain possible).

SECONDARY OUTCOMES:
The Benefit, Satisfaction, and Willingness to Continue of each participant after the procedure | 2 weeks +/- 7 days after procedure and 3 +/- 7 days months after procedure
  The Benefit, Satisfaction, and Willingness to Continue (BSW) questionnaire is a validated instrument administered by the physician. It asks participants if they had benefit, satisfaction, and a willingness to continue from a specific treatment. If yes, responses range from 1(little benefit, little, satisfaction, a little bit willing) to 2(much benefit, very satisfied, very willing).
Change in extent of Overactive Bladder Symptoms before and after receiving the procedure | Pre procedure, 2 weeks +/- 7 days after procedure, and 3 +/- 7 days months after procedure
  The Overactive Bladder questionnaire (OAB-q) short form is a validated instrument that measures the extent to which participants have various symptoms of OAB over the past 4 weeks. The responses range from 1(not at all) to 6(a very great deal).
The Prevalence of complications with botox after receiving the procedure | 2 weeks +/- 7 days after procedure, and 3 +/- 7 days months after procedure
  The Complications with Botox survey is an instrument used to measure if and how many times participants experienced UTIs, difficulty urinating, or hematuria after the Botox procedure. Participants self-report the number of times if they have experienced the side effect.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Lanzer, MD, Principal Investigator — Augusta University; Emily Grandprey, DO, Study Director — Augusta University; Emily Lluch, Study Director — Augusta University; Ahana Gaurav, Study Director — Augusta University

IPD SHARING:
Plan to Share IPD: No